CLINICAL TRIAL: NCT00104039
Title: Investigating the Neuro-Cognitive Underpinnings of the Emotional Dysfunction Linked to Childhood Behavioral Disturbance
Brief Title: Brain Changes in Children and Adolescents With Behavioral Problems
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050105; 05-M-0105
Record Dates: First submitted 2005-02-19; First posted 2005-02-21 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2016-07-21

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Mental Disorders Diagnosed in Childhood; Conduct Disorder
Keywords: Amygdala; Orbital Frontal Cortex; Serotonin; Orbitofrontal Cortex; Attention Deficit Hyperactivity Disorder; ADHD; Anti-Social Behavior; Healthy Volunteer; HV
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Conduct Disorder; Antisocial Personality Disorder

SUMMARY:
Purpose:

This study will examine brain activity in children age 10-18 with disruptive behavior problems, including conduct disorder (CD), oppositional defiant disorder (ODD), and attention deficit hyperactivity disorder (ADHD), compared with children without behavioral problems. Our goal is to examine differences in how emotions, social situations, and problem-solving situations are processed in the brain across these groups of children.

DETAILED DESCRIPTION:
OBJECTIVE:

The goal of this protocol is to investigate the neuro-cognitive underpinnings of the emotional dysfunction linked to childhood behavioral disturbance; in particular, Conduct Disorder with elevated callous-unemotional (CU) traits (CD+CU), Conduct Disorder with non elevated CU traits (CD-CU), but also ADHD. The functional hypotheses that we are testing with both neuro-cognitive and neuro-imaging paradigms are that: (1) CD+CU, but not ADHD, is associated with dysfunction in the formation and operational use of stimulus-punishment and, to a lesser extent, stimulus-reward association information; (2) CD-CU is associated with heightened threat sensitivity and impairment in executive systems involved in emotional regulation; and (3) that ADHD and CD-CU, is associated with impairment in executive systems related to the representation and execution of task demands.

STUDY POPULATION:

160 children with Conduct Disorder (CD) and high CU traits (the CD+CU group); 160 children with CD and low CU traits (the CD-CU group); 160 children with ADHD; and 160 healthy volunteer children. All children will be between the ages of 10 and 17. Both males and females will be enrolled.

DESIGN:

The current study will have two phases: i) neuropsychological assessment and training in an MRI simulator (up to 4 hours); ii) The MRI scanning session (up to 2 hours, no more than 90 minutes in scanner). Participants, if they are willing, may be invited to participate in more than one scanning session (up to a maximum of 3 120 minute sessions) or neuro-cognitive testing session.

OUTCOME MEASURES:

Behaviorally, we predict that children with CD+CU and children with CD-CU will present with impairment on tasks that involve either the formation or operational use of particular stimulus-punishment associations (e.g., the subjective value learning task and emotional interrupt task). However, the nature of this impairment with be qualitatively different. For example, we predict that youth with CD+CU will show reduced interference by emotional distracters on the emotional interrupt task but that youth with CD-CU will show decreased interference. In contrast, we predict that children with ADHD, but no CD, will show no behavioral impairment on such tasks. However, we predict that children with ADHD and children with CD-CU will present with impairments on executive function tasks (e.g., the Number Stroop paradigm). In contrast, we predict that children with CD+CU will show no impairment on these tasks. At the anatomical level, we anticipate reduced activation of emotional related systems in children with CD+CU, but increased activation in children with CD-CU, during emotional impact tasks (in particular, reduced activation of the amygdala, regions of orbitofrontal cortex and anterior cingulate). We anticipate that the neural response of children with ADHD during these tasks will be less anomalous. We anticipate that the neural response of children with ADHD and children with CD-CU during the performance of response control tasks to be anomalous (with considerable greater recruitment of anterior and posterior compensatory systems).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Individuals with CD + CU: Male and female subjects aged 8-18 who score equal to or more than 20 on the APSD/PCL-YV. Children with antisocial behavioral problems on medications with psychotropic effects will be considered if their target behaviors persist despite the use of medications. In these children, only simple stimulant medications will be held for 48 hours. These include methylphenidate, amphetamine and their derivatives including Ritalin, Ritalin SR, Ritalin LA, Methylin, Methlin ER, Metadate CD, Concerta, Dexedrine, Dextrostat, Dexedrine Spansule, Adderall, Adderall XR, and Focalin. Medications like Strattera (atomoxetine), bupropion (Wellbutrin), modafinil (Provigil), or valproic acid (Depakote), or other mood stabilizers are not safe to stop suddenly and children taking these medications will not be asked to stop them.
  2. Individuals with CD-CU: Male and female subjects aged 8 -18 who score less than 20 on the APSD/PCL-YV. Children with antisocial behavioral problems on medications with psychotopic effects will be considered if their target behaviors persist despite the use of medications. In these children, only simple stimulant medications will be held for 48 hours. These include methylphenidate, amphetamine and their derivatives including Ritalin, Ritalin SR, Ritalin LA, Methylin, Methlin ER, Metadate-CD, Concerta, Dexedrine, Dextrostat, Dexedrine Spansule, Adderall, Adderall XR, and Focalin Medications like Starattera (atomoxetine), bupropion (Wellbutrin), modafinil (Provigil), or valproic acid (Depakote), or other mood stabilizers are not safe to stop suddenly and children taking these medications will not be asked to stop them.
  3. Individuals with ADHD: Male and female subjects aged 8-18 who currently meet DSM-IV criteria for ADHD. The diagnosis will be made on the basis of a K-SADS-PL interview with the parent and a t score >65 on the hyperactivity-impulsivity subscale of the Connors Teacher Scale. Participants in this group will have APSD scores <20.
  4. Comparison individuals: Male and female subjects aged 8-18 who are free from any current or past psychopathology (all will score less than 20 on the APSD/PCL-YV).

EXCLUSION CRITERIA:

1. I.Q.< 75.
2. Ongoing medical illness other than those listed in the inclusion criteria for the respective groups that require use of any medication that may have psychotropic effects. For example, a patient with history of mild asthma that did not require medication may be included, however a patient with asthma requiring use of beta blockers, steroids, etc. would not be included. For children with ADHD or healthy volunteer children, a contraindication to discontinuing medication for 48 hours. Only simple stimulant medications will be held for 48 hours. These include methylphenidate, amphetamine and their derivative including Ritalin, Ritalin SR, Ritalin LA, Methylin, Methlin ER, Metadate CD, Concerta, Dexedrine, Dextrostat, Dexedrine Spansule, Adderall, Adderall XR, and Focalin. Medications like Strattera (atomoxetine), bupropion (Wellbutrin), or modafinil (Provigil) are not safe to stop suddenly and children with ADHD taking these medications will not be included.
3. Subjects with psychopathic tendencies who receive a diagnosis of an anxiety or mood disorder as determined by a clinical and K-SAD review conducted by a psychiatrist will be excluded. Additionally, children with active psychosis, pervasive developmental disorders or Tourette s syndrome will be excluded.
4. Children with CD-CU will be evaluated through the KSAD and clinical review by a psychiatrist. Explicit exclusions include active psychosis, Pervasive Developmental Disorders and Tourette s syndrome. Children with anxiety disorders will be included given the high comorbidity of CD-CU and anxiety disorders.
5. Individuals with ADHD will be evaluated through the KSAD and clinical review by a psychiatrist. Those children who receive diagnosis of mood disorders through this evaluation process will be excluded. Additional explicit exclusions include active psychosis, Pervasive Developmental Disorders and Tourette s syndrome. Children with anxiety disorders will be included given the high comorbidity of ADHD and anxiety disorders.
6. Any other psychiatric disorder that is sufficiently severe to require specific treatment, with the exception of those listed in the inclusion criteria for the respective groups.
7. Neurologic disorder (including seizures).
8. Any metallic objects in the body. Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
9. Claustrophobia: participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2005-02-17; Study Completion 2016-07-21

CONTACTS AND LOCATIONS:
Overall Officials: James J Blair, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ambrogi Lorenzini CG, Baldi E, Bucherelli C, Sacchetti B, Tassoni G. Neural topography and chronology of memory consolidation: a review of functional inactivation findings. Neurobiol Learn Mem. 1999 Jan;71(1):1-18. doi: 10.1006/nlme.1998.3865. PMID 9889069
- [Background] Aron AR, Fletcher PC, Bullmore ET, Sahakian BJ, Robbins TW. Stop-signal inhibition disrupted by damage to right inferior frontal gyrus in humans. Nat Neurosci. 2003 Feb;6(2):115-6. doi: 10.1038/nn1003. No abstract available. PMID 12536210
- [Background] Babinski LM, Hartsough CS, Lambert NM. Childhood conduct problems, hyperactivity-impulsivity, and inattention as predictors of adult criminal activity. J Child Psychol Psychiatry. 1999 Mar;40(3):347-55. PMID 10190336
- [Derived] Hwang S, Meffert H, Parsley I, Tyler PM, Erway AK, Botkin ML, Pope K, Blair RJR. Segregating sustained attention from response inhibition in ADHD: An fMRI study. Neuroimage Clin. 2019;21:101677. doi: 10.1016/j.nicl.2019.101677. Epub 2019 Jan 15. PMID 30682530
- [Derived] Tyler PM, White SF, Thompson RW, Blair RJR. Applying a Cognitive Neuroscience Perspective to Disruptive Behavior Disorders: Implications for Schools. Dev Neuropsychol. 2019 Jan-Feb;44(1):17-42. doi: 10.1080/87565641.2017.1334782. Epub 2018 Feb 12. PMID 29432037
- [Derived] White SF, Thornton LC, Leshin J, Clanton R, Sinclair S, Coker-Appiah D, Meffert H, Hwang S, Blair JR. Looming Threats and Animacy: Reduced Responsiveness in Youth with Disrupted Behavior Disorders. J Abnorm Child Psychol. 2018 May;46(4):741-754. doi: 10.1007/s10802-017-0335-0. PMID 28776147
- [Derived] White SF, VanTieghem M, Brislin SJ, Sypher I, Sinclair S, Pine DS, Hwang S, Blair RJ. Neural Correlates of the Propensity for Retaliatory Behavior in Youths With Disruptive Behavior Disorders. Am J Psychiatry. 2016 Mar 1;173(3):282-90. doi: 10.1176/appi.ajp.2015.15020250. Epub 2015 Oct 6. PMID 26441155